CLINICAL TRIAL: NCT04889638
Title: Comprehensive Tobacco Cessation for Residents of Baltimore City Public Housing
Brief Title: Tobacco Cessation in Public Housing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); Community Partnership and Collaboration Core Pilot Grant (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00224186; UL1TR003098 (NIH)
Record Dates: First submitted 2021-05-12; First posted 2021-05-17 (Actual); Results first posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Smoking Cessation; Smoking Reduction; Smoking, Tobacco
MeSH Terms: conditions — Smoking Cessation; Smoking Reduction; Tobacco Smoking

STUDY DESIGN:
Intervention Model Description: Pre-post study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cessation intervention (Experimental): Participants will undergo pre-/post-comparisons of a personalized, remote smoking cessation intervention composed of two main elements: a) prescription and monitoring of nicotine (e.g., replacement therapy) and/or non-nicotine pharmacotherapies (e.g., varenicline) and b) cessation-centered motivational messaging.
  Interventions: Other: Cessation Intervention

INTERVENTIONS:
Other: Cessation Intervention — 1. Pharmacotherapy selection, prescription and monitoring of up to two types of cessation pharmacotherapies: Nicotine replacement therapy (gum, lozenge and transdermal patch) and non-nicotine replacement therapy (varenicline).
  2. Remote video-conferencing and mobile phone-based, personalized motivational messaging

SUMMARY:
The inequity in cessation resources is at forefront in the recently enacted nationwide smoking ban in public housing facilities. The critical component lacking from the federal decree was a practical smoking cessation strategy to address the real-world needs of active smokers who maintain cigarette usage. The investigator's proposal is ideally situated for this contemporary moment when low-income smokers in public housing are signing leases describing the potential for smoking-related evictions and thus at least contemplating smoking modification. The investigator's project is centered around the residents of Baltimore City Public Housing which is among the larger-sized U.S. public housing agencies. Using a human-centered design (HCD) approach, the investigators are refining and testing a community-centric cessation strategy defined by two core elements: a) durable and jointly linked community/hospital infrastructure systems (remote cessation specialist staffing and drug supplies) and strong on-site (public housing) residential leadership commitment to cessation improvement. These dual features, along with adaptable elements that can be modified to a variety of local/national housing settings, defines how the investigator's project will overcome the implementation gaps defining failed smoking cessation efforts in lower-income settings. The objective of this project is to test the feasibility of the intervention package among local housing contextual factors that could impact both the acceptability and adoptability of the investigator's project. Using a collection of formative and implementation evaluation measures, the investigator's academic-community partnership project is well positioned to create an adaptable and customizable intervention that can be scaled in similar housing populations.

DETAILED DESCRIPTION:
Lower socioeconomic populations continue to remain at high risk for tobacco use and suffer disproportionately from tobacco-related disease. Evidence is lacking of ways to optimally deliver behavioral and pharmaceutical-based cigarette smoking cessation interventions in real-world environments among disadvantaged cohorts where geographic, socioeconomic and technological disparities often undermine the effectiveness of evidence-based smoking cessation efforts. The investigator's study focuses on residents of public housing in Baltimore City, a population who face multiple socioeconomic stressors and of whom up to 1/3 are assumed conventional cigarette users.

The investigator's project uses a partnership between the Housing Authority of Baltimore City (HABC) and Johns Hopkins School of Medicine to enact a remote (off-site) cessation program in two public housing complexes under the management of HABC. The investigator's program will institute evidence-based practices in an accessible manner for the residents at both sites. The investigator's program's key features include the remote recruitment, prescription, delivery and management of evidence-based nicotine pharmacotherapies, and provision of cessation counseling.

To assess the feasibility of study design, the investigator's project specifically focuses on the following eight elements: a) recruitment of smokers expressing a motivation to reduce or quit smoking, b) Consent process, c) nicotine and non-nicotine pharmacotherapy selection, screening, prescription, delivery, storage management (participation education, side-effecting monitoring), and return of unused drug supplies, d) Administration and perceived utility of motivational interviewing regarding smoking reduction and cessation, e) Delivery of study reimbursement, f) Utility of weekly text reminders of study participation and final endpoint, g) acceptability of outcome measures, h) acceptability and evaluation of joint project oversight with community stakeholders.

The project will enroll eighty participants to determine feasibility endpoints. All participants will receive the intervention, as preferred by community partners. Participants will serve as the participants own control, which in turn means that the investigators will compare the intervention's effect at an individual level. All participants will be offered over a 4-week period both a long-acting nicotine controller medication (varenicline or nicotine patch) and short-acting medication to address acute urges to smoke (nicotine gum/lozenge). Each week participants will be monitored and receive cessation-directed counseling. If medication questions or concerns arise, patients will have access to 24-hour phone support. The results of the project will be reviewed with participants, community partners and academic team.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age to 99 years old
* Self-reported smoker with either daily or weekly cigarette use, as well as expressed desire to reduce or quit smoking
* Proof of residence at Douglass or Brooklyn Homes through verbal acknowledgement by the Service Coordinators at each of the public housing sites.
* Working cell phone with ability to text for the duration of the study
* Active health insurance (for pharmacotherapy billing)

Exclusion Criteria:

* Pregnant - women will verbally acknowledge that they are not pregnant
* Breastfeeding - women who are verbally acknowledge they are breastfeeding will be excluded from the study.
* Ongoing participation in a tobacco cessation program or related tobacco intervention study
* Unable to verbally state that they are willing to reduce or quit smoking upon recruitment and screening
* Adults lacking capacity to consent
* Non-English speakers
* Self-reported usage of only non-combustible tobacco products, such as smokeless tobacco or Electronic Nicotine Delivery Devices (ENDS).
* Anticipated relocation outside of Douglass or Brooklyn Homes prior to the final study visit

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2024-04-03 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Panagis Galiatsatos, Principal Investigator — Johns Hopkins University
Locations (1):
- Creative Alternative, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 2 participating housing units.
Groups:
- Recruitment Arm: Each participant was expected to commit to a 4-week study that will be administered both in-person at their housing site and remotely. Remote study visits will occurred by either a video conference call or standard audio phone call. At each session, the following 2 things were discussed: Drug education, proper drug usage and side-effect monitoring of a 4-week supply of nicotine medications that are delivered to participant's home address prior to starting the first study visit.
  Motivational counseling to help you quit or reduce smoking.
Period: Overall Study
Arm/Group | Recruitment Arm
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cessation Intervention
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 18
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
PROMIS Nicotine Dependence Survey Score [Mean (Standard Deviation); unit: score on a scale] — The scores range from 8 - 40. The lower end of the range indicates no nicotine dependence and the upper end of the range correlates with a high degree of dependence.
  score on a scale | 25.3 (6.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Nicotine Dependence (Short Form 8a) Score
Description: This outcome measures assesses cravings or withdrawal that occurs upon brief cessation of smoking, smoking temptations, compulsive use, and tolerance.
  The scores range from 8 - 40. The lower end of the range indicates no nicotine dependence and the upper end of the range correlates with a high degree of dependence.
Time Frame: Baseline, 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cessation Intervention
Number analyzed (Participants) | 18
score on a scale | 11.2 (6.5)

2. Secondary Outcome: Change in PROMIS Coping Expectancies (Short Form 4a) Score
Description: This outcome measure assesses smokers' tendency to use smoking as a means of coping with negative affect and stress.
  The scores range from 4 - 20. A score of 4 indicates cigarettes are not being used to cope with life experience and mental health; a maximum of 20 indicates cigarettes are being used always or very much to address both negative life experiences and mental health.
Time Frame: Baseline, 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cessation Intervention
Number analyzed (Participants) | 18
score on a scale | 5.2 (3.1)

3. Secondary Outcome: Change in PROMIS Emotional and Sensory Expectancies (Short Form 6a) Score
Description: This outcome measure assesses perceptions of improved cognitive abilities, positive affective states, and pleasurable sensorimotor sensations due to smoking.
  The scores range from 6 - 30. A score of 6 indicates cigarettes are not being used to enhance emotional and sensory experiences; a maximum of 30 indicates cigarettes are strongly (or very much) used to improve both emotional and sensory experiences.
Time Frame: Baseline, 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cessation Intervention
Number analyzed (Participants) | 18
score on a scale | 7.1 (2.3)

4. Secondary Outcome: Change in PROMIS Health Expectancies (Short Form 6a) Score
Description: This outcome measure assesses perceptions of improved cognitive abilities, positive affective states, and pleasurable sensorimotor sensations due to smoking.
  The scores range from 6 - 30. A score of 6 indicates smoking cigarettes are not perceived at all as being associated with negative health experiences, including changes in cognition, affect and sensorimotor sensations; a score of 30 translates to a perception that cognition, affect and sensorimotor sensations are very much associated with smoking.
Time Frame: Baseline, 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cessation Intervention
Number analyzed (Participants) | 18
score on a scale | 6.3 (2.5)

5. Secondary Outcome: Change in PROMIS Psychosocial Expectancies (Short Form 6a) Score
Description: This outcome measure assesses smokers' beliefs about aspects of social disapproval and disappointment in oneself that are experienced as a result of smoking.
  The scores range from 6 - 30. A score of 6 indicates smoking cigarettes are not perceived at all as being associated with social disapproval and disappointment in oneself; a score of 30 translates to a perception that smoking is very much associated with social disapproval and disappointment in oneself
Time Frame: Baseline, 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cessation Intervention
Number analyzed (Participants) | 18
score on a scale | 5.1 (2.2)

6. Secondary Outcome: Change in PROMIS Social Motivations (Short Form 4a) Score
Description: This outcome measure assesses smokers' assesses self-reported social factors that influence smoking behavior.
  The range of scores is from 4 - 20. A score of 4 indicates there is not any perceived association between smoking and social factors; a score of 20 indicates a very strong perception that smoking is associated with social factors.
Time Frame: Baseline, 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cessation Intervention
Number analyzed (Participants) | 18
score on a scale | 7.3 (4.3)

ADVERSE EVENTS:
Time Frame: Up to 6-months
Groups:
- Cessation Intervention: Participants will undergo pre-/post-comparisons of a personalized, remote smoking cessation intervention composed of two main elements: a) prescription and monitoring of nicotine (e.g., replacement therapy) and/or non-nicotine pharmacotherapies (e.g., varenicline) and b) cessation-centered motivational messaging.
  Cessation Intervention: 1. Pharmacotherapy selection, prescription and monitoring of up to two types of cessation pharmacotherapies: Nicotine replacement therapy (gum, lozenge and transdermal patch) and non-nicotine replacement therapy (varenicline).
  2. Remote video-conferencing and mobile phone-based, personalized motivational messaging
Arm/Group | Cessation Intervention
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-10): https://cdn.clinicaltrials.gov/large-docs/38/NCT04889638/Prot_SAP_000.pdf
  • Informed Consent Form (2024-02-27): https://cdn.clinicaltrials.gov/large-docs/38/NCT04889638/ICF_001.pdf